CLINICAL TRIAL: NCT03296514
Title: Mindfulness-Based Stress Reduction Study for Couples
Brief Title: Mindfulness Based Stress Reduction for Metabolic Syndrome
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Joan Monin, Associate professor with term, Yale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2000020175
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control (No Intervention): Will receive voucher for MBSR after study is concluded
- Intervention (Other): These people will receive the MBSR
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Eight week class on MBSR in addition to an orientation class and a half day retreat
  Arms: Intervention

SUMMARY:
Mindfulness based stress reduction offered to couples where one has metabolic syndrome to see if their stress is reduced as measured by bio markers and surveys

DETAILED DESCRIPTION:
This is a pilot study being designed to pilot a MBSR program for the purposes of future research.The investigators will be using two cohorts. One who will get the intervention and the other who will be wait listed and receive the intervention at a later date. Eight week mindfulness class offered to couples, who also attend an orientation session and a half day retreat with other couples to learn how to control stress through mindfulness meditation practices. Participants will come for lab work before intervention, eight weeks after initial class and at the end of entire program. Bio- markers to be measured are waist circumference, FBS and cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Participant has 3 of the following: a Abdominal Obesity; b. Hypertriglyceridemia; c. Low High Density Lipoproteins (HDL); d. High Blood Pressure; e. High Fasting Blood Sugar (FBS)
* Participant must be married or co- habituating
* Both partners are over sixty

Exclusion Criteria:

* Either partner is non- English speaking
* Either partner practices mind- body therapies more than once a week/
* Either partner taking psychiatric medicine

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Self- reported physical health status | Up to three weeks after intervention ends
  SF 12
Perceived stress | Up to three weeks after intervention ends
  Perceived stress scale,
Mindfulness Skills | Up to three weeks after intervention ends
  Kentucky Inventory of Mindfulness Skills

CONTACTS AND LOCATIONS:
Overall Officials: Joan Monin, PhD, Principal Investigator — Professor
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gu J, Strauss C, Bond R, Cavanagh K. How do mindfulness-based cognitive therapy and mindfulness-based stress reduction improve mental health and wellbeing? A systematic review and meta-analysis of mediation studies. Clin Psychol Rev. 2015 Apr;37:1-12. doi: 10.1016/j.cpr.2015.01.006. Epub 2015 Jan 31. PMID 25689576
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Background] Creswell JD, Myers HF, Cole SW, Irwin MR. Mindfulness meditation training effects on CD4+ T lymphocytes in HIV-1 infected adults: a small randomized controlled trial. Brain Behav Immun. 2009 Feb;23(2):184-8. doi: 10.1016/j.bbi.2008.07.004. Epub 2008 Jul 19. PMID 18678242
- [Background] Creswell JD, Irwin MR, Burklund LJ, Lieberman MD, Arevalo JM, Ma J, Breen EC, Cole SW. Mindfulness-Based Stress Reduction training reduces loneliness and pro-inflammatory gene expression in older adults: a small randomized controlled trial. Brain Behav Immun. 2012 Oct;26(7):1095-101. doi: 10.1016/j.bbi.2012.07.006. Epub 2012 Jul 20. PMID 22820409
- [Background] Cramer H, Haller H, Lauche R, Dobos G. Mindfulness-based stress reduction for low back pain. A systematic review. BMC Complement Altern Med. 2012 Sep 25;12:162. doi: 10.1186/1472-6882-12-162. PMID 23009599
- [Background] Biegel GM, Brown KW, Shapiro SL, Schubert CM. Mindfulness-based stress reduction for the treatment of adolescent psychiatric outpatients: A randomized clinical trial. J Consult Clin Psychol. 2009 Oct;77(5):855-66. doi: 10.1037/a0016241. PMID 19803566
- [Background] Birnie K, Garland SN, Carlson LE. Psychological benefits for cancer patients and their partners participating in mindfulness-based stress reduction (MBSR). Psychooncology. 2010 Sep;19(9):1004-9. doi: 10.1002/pon.1651. PMID 19918956

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03296514/Prot_000.pdf
  • Informed Consent Form (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT03296514/ICF_001.pdf